CLINICAL TRIAL: NCT05929300
Title: Developing and Pilot-testing a Yoga Program to Address Post-prostatectomy Side-effects Among Veterans With Prostate Cancer
Brief Title: A Yoga Program for Patients Undergoing Prostate Cancer Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PPO 21-225
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer; Erectile Dysfunction; Urinary Incontinence
Keywords: Yoga
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction; Urinary Incontinence | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The study design entails randomizing ~34 Veterans who are undergoing radical prostatectomy (RP) for prostate cancer (PCa) to either usual care or a twice-weekly hybrid (in-person and virtual) yoga program that includes up to 4 weeks of pre-habilitation yoga and 8 weeks of post-RP yoga. Participants will provide data at three time points: baseline/pre-yoga (T1), completion of~ 4 weeks of pre-RP yoga (T2), and completion of 8 weeks of post-RP yoga (T3). Veterans randomized to the intervention will be asked to routinely practice yoga (at least 15 min/day). The control group will consist of "usual care" patients. It is current practice for all patients to: 1) receive a handout that covers Kegel exercises; and, 2) instruction from a nurse who teaches the patient how to perform the exercises. There is no referral to a physical therapist unless progression indicates a need for it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga (Experimental): The study design entails randomizing ~34 Veterans who are undergoing RP for PCa to either usual care or a twice-weekly hybrid (in-person and virtual) yoga program that includes up to 4 weeks of pre-habilitation yoga and 8 weeks of post-RP yoga. Participants will provide data at three time points: baseline/pre-yoga (T1), completion of~ 4 weeks of pre-RP yoga (T2), and completion of 8 weeks of post-RP yoga (T3). Data collection for the control group will parallel that of the yoga group. Times of data collection are consistent with other yoga trials. Veterans randomized to the intervention will be asked to routinely practice yoga (at least 15 min/day).
  Interventions: Behavioral: Yoga; Other: Usual Care
- Usual Care (Active Comparator): The control group will consist of "usual care" patients. It is current practice for all patients to: 1) receive a handout that covers Kegel exercises; and, 2) instruction from a nurse who teaches the patient how to perform the exercises. There is no referral to a physical therapist unless progression indicates a need for it.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Yoga — The yoga program includes up to 4 weeks of pre-habilitation yoga and 8 weeks of post-surgery yoga. The yoga program includes basic yoga poses and breathing exercises.
  Arms: Yoga
Other: Usual Care — This consists of "usual care" patients. It is current practice for all patients to: 1) receive a handout that covers Kegel exercises; and, 2) instruction from a nurse who teaches the patient how to perform the exercises. There is no referral to a physical therapist unless progression indicates a need for it.

SUMMARY:
Men with localized prostate cancer (PCa) are often treated with surgery, a treatment that is associated with high rates of side effects such as erectile dysfunction (ED) and urinary incontinence (UI) which impact quality of life. Yoga may improve control of UI and improve ED by bringing awareness to and strengthening the pelvic floor musculature. The randomized controlled pilot study is to assess the feasibility of an innovative hybrid (in-person and virtual) twice-weekly yoga program that includes a prehabilitation component and to obtain preliminary data that will help assess its potential effectiveness in alleviating PCa treatment symptom burden (primarily ED and UI). The long-term goal is to develop a scalable and sustainable yoga program that helps cancer survivors manage their treatment side effects.

DETAILED DESCRIPTION:
Those who are treated with radical prostatectomy (RP) for prostate cancer (PCa) often experience side effects including erectile dysfunction (ED) and urinary incontinence (UI). The side effects of treatment often persist for years and can contribute to anxiety and depression. Yoga, which includes breath work, meditation, and physical poses, may be an effective intervention for treating side effects of RP. To facilitate uptake and maximize its effectiveness, the investigators are initiating the intervention prior to surgery (prehabilitation) and delivering it using a blended approach (i.e., in-person and online sessions).

The proposed intervention is innovative in several ways. First, it applies yoga to a relatively new patient population (men with PCa) and sets of outcomes (ED and UI). Second, the intervention is being tailored to the patient and delivered using a blended model. The first session is in-person and used to tailor the yoga poses according to a Veteran's comfort and ability. Subsequent sessions will take place online alongside ongoing patient cohorts. Third, the intervention includes a prehabilitation component that aims to further dampen the side effects of RP.

The long-term goal of this research is to optimize the QoL and patient experience for men with PCa. To that end, the investigators seek to assess the feasibility of an innovative blended (in-person and online) yoga program and to obtain preliminary data on its potential effectiveness in alleviating PCa treatment symptom burden. The specific aims are to: 1) determine the feasibility (including demand, safety and acceptability) of the intervention for men receiving a radical prostatectomy; and 2) obtain preliminary data to estimate the potential impact of the intervention on ED and UI (primary outcomes), well-being (e.g., cancer fatigue, stress, anxiety), and QoL. Methodology: For this pilot study, 34 Veterans who are undergoing a radical prostatectomy for PCa treatment will be randomized to either the intervention or standard of care. The intervention is a blended twice-weekly yoga program that includes a prehabilitation phase. ED and UI (primary outcomes) as well as mental health well-being (e.g. stress, anxiety), including QoL (secondary outcomes). Program uptake and attrition will be tracked and compared between groups. Baseline and follow-up data on outcomes will be collected via survey. Safety will be closely monitored. Veterans' experiences with and perceptions of the program will be assessed through a post-intervention survey.

ELIGIBILITY:
Inclusion Criteria:

* patients must be age 18 year or older
* have a biopsy-proven diagnosis of localized prostate cancer
* scheduled to undergo robotic-assisted or open radical prostatectomy
* speak English
* willing and able to attend an in-person yoga session at Hines VA
* possess hardware and internet connectivity that will enable participation in virtual yoga classes

Exclusion Criteria:

* patients will be excluded if currently participating in yoga practice (twice weekly in past three months) and have any of the following conditions:

  * neurogenic bladder
  * (uncontrolled/major) cardiac arrhythmia
  * psychosis
  * cognitive impairment
* patients will be excluded if they are planning to move outside of the Chicago area
* unable to participate in low- to moderate-intensity physical activity
* currently experiencing issues around substance abuse (not including prescription opioids)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Change in level of erectile dysfunction from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  The 5-item International Index of Erectile Function diagnostic tool was developed in consultation with an international panel of experts for use in determining treatment efficacy in clinical trials. The scores range from 0 to 25 with scores >21 indicating normal erectile function.
Change in level of urinary incontinence from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  The 4-item International Consultation on Incontinence Questionnaire-Urinary Incontinence assesses symptoms of incontinence with higher scores indicating more severe symptoms. The scores range from 0 to 21 with scores>9 depicting very severe impact on daily life activities.

SECONDARY OUTCOMES:
Change in level of cancer-related fatigue from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  The 9-item Brief Fatigue Inventory questionnaire can assess fatigue severity. Each item ranges from 0-10 with values >7 denoting severe interference with daily life activities.
depression | Change in level of depression from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga
  The Patient Health Questionnaire (PHQ-9) provides a brief measure of depression severity (i.e., mild, moderate, moderately severe, and severe) over the past two weeks. The scores range from 0 to 27 with scores>19 depicting severe depression.
Change in level of anxiety from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  The Generalized Anxiety Disorder 7-item instrument (GAD-7) measures the level of anxiety with a score of 10 or more (out of a total score of 21) indicating clinically significant anxiety.
Change in level of stress from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  The Perceived Stressor Scale is a 10-item questionnaire that assesses the degree to which one finds life unpredictable, uncontrollable or overloaded over the past month. The scores range from 0 to 40 with scores>26 depicting high perceived stress.
Change in level of quality of life from baseline to 4-weeks of pre-habilitation yoga and to 8-weeks of rehabilitation yoga | Through study completion, an average of 16 weeks
  Quality of life will be evaluated via the Functional Assessment of Cancer Therapy questionnaire for patients with PCa (FACT-P). Total scores range from 0 to 104 with higher scores denoting higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Silva, PhD MPH BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
We will use the Safe Harbor Method to de-identify the data set include a limited set of the most relevant variables to help ensure that patient confidentiality and privacy is maintained. The VHA privacy officer will certify whether the data set meet conditions for disclosure to the public. Final data sets will be maintained locally. Guidance on request and distribution processes will be provided by Office of Research and Development. Data users will have to sign a Data Use Agreement in compliance with privacy regulations.
Supporting Information: Study Protocol, SAP, ICF